CLINICAL TRIAL: NCT04837456
Title: First Affilated Hospital of Jinzhou Medical University
Brief Title: Metabolic Syndrome and Degenerate Meniscus Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Jingzhou (Other)
Responsible Party: Principal Investigator, Hongyu Wang, chief residents, The First People's Hospital of Jingzhou
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FirstJingzhou
Record Dates: First submitted 2021-03-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Syndrome; Meniscus; Degeneration
Keywords: Metabolic Syndrome; degenerate meniscus lesions; Calorie restricted diet; exercise; arthroscopic partial meniscectomy
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calorie restricted diet and excecise intervention (Experimental): a balanced diet that provided an energy deficit of 800 kcal/day from their daily energy requirement [36]. Macronutrient content of low caloric diet, expressed as percentage of ingested energy with carbohydrates 45-65%; fat 20-35%; and protein 10- 35%[36].Each session was approximately 150 minutes one week for six months and consisted of aerobic exercises, resistance training, and exercises to improve flexibility and balance.
  Interventions: Dietary Supplement: Calorie restricted diet and exercise intervention
- libitum diet and waiting list control group (Experimental): participants then underwent a calorie of 2000 calorie above based on libitum free diets recommended to adults and normal physical activity without exercise during the program.
  Interventions: Procedure: libitum diet and waiting list control group
- Early APM group (Experimental): Early APM group participants received APM with syndrome within 3 to 6 months
  Interventions: Procedure: Early arthroscopic partial menisectomy group
- delayed APM group recruit participants with symptoms lasting for more than 6 months (Experimental): delayed APM group recruit participants with symptoms lasting for more than 6 months
  Interventions: Procedure: delayed APM group recruit participants with symptoms lasting for more than 6 months

INTERVENTIONS:
Dietary Supplement: Calorie restricted diet and exercise intervention — the calorie restricted diet were prescribed a balanced diet that provided an energy deficit of 800 kcal/day from their daily energy requirement.Macronutrient content of low caloric diet, expressed as percentage of ingested energy with carbohydrates 45-65%; fat 20-35%; and protein 10- 35%[36]. Participants were guided by a dietitian for adjustments of their caloric intake weekly for six months.Participants performed 1 or 2 sets at a resistance of approximately 65% of their one-repetition maximum, with 8 to 12 repetitions of each exercise; they gradually increased the intensity to 2 to 3 sets at a resistance of approximately 80% of their one-repetition maximum, with 6 to 8 repetitions of each exercise.
  Arms: Calorie restricted diet and excecise intervention
Procedure: libitum diet and waiting list control group — libitum diet and waiting list control group, participants then underwent a calorie of 2000 calorie above based on libitum free diets recommended to adults and normal physical activity without exercise during the program.
  Arms: libitum diet and waiting list control group
Procedure: Early arthroscopic partial menisectomy group — Early APM group participants received APM with syndrome within 3 to 6 months
  Arms: Early APM group
Procedure: delayed APM group recruit participants with symptoms lasting for more than 6 months — delayed APM group recruit participants with symptoms lasting for more than 6 months
  Arms: delayed APM group recruit participants with symptoms lasting for more than 6 months

SUMMARY:
The aim is to determine the outcomes of calorie-restricted diet and exercise intervention; libitum diet and waiting list control; early arthroscopic partial meniscectomy(APM) or delayed APM effect on MetS patients with Degenerate menisucus lesions.

DETAILED DESCRIPTION:
The investigators recruited 180 patients with Metabolic Syndrome and knee symptoms with degenerate meniscus lesions by MRI from orthopaedics department from June 2017 to March 2020 at First Affiliated Hospital of Jinzhou Medical University. Participants were diagnosed with MetS and degenerate meniscus tear with a mild or no osteoarthritis KL<2 verified by X ray. Participants were randomly dividied into calorie-restricted diet and exercise intervention group; libitum diet and waiting list control group; early APM (syndrome within 3-6 months) group or a delayed APM(syndrome more than 6 months) group as a computer sequenced number. The primary outcome was the change in metabolic syndrome components and knee function score of WOMAC, KOOS,WOMET,IKDC were determined by two fixed orthopadic surgeons who were blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be age between 35 and 70 years old;
* Clinical diagnosis of metabolic syndrome;
* Clinical diagnosis of 3 grade degneration meniscus leisons;

Exclusion Criteria:

* Must be able to have no acute knee injury such as car crash or acute sports injury;
* Must be able to have no knee surgeries history;
* Must be able to have no rheumatoid arthritis or serious knee osteoarthritis with deformity;
* Must be able to have no contraindications to MRI;
* Must be able to have no severe cardiopulmonary disease;
* Must be able to have no musculoskeletal or neuromuscular impairments ;
* Must be able to have good visual, hearing, or cognitive;

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 189 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Knee KOOS4 | up to 12 months
  the Knee injury and Osteoarthritis Outcome Score (KOOS) holds five subscales: (1) Pain (9 items); (2) other Symptoms (7 items); (3) Activities of Daily Living (ADL, 17 items); (4) Sport and Recreation function (Sport/Rec, 5 items); and (5) knee-related Quality of Life (QoL, 4 items). Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems) life (KOOs 4 ) were assessed.One of the most frequently-used knee-specific PROMs is the Knee injury and Osteoarthritis Outcome Score (KOOS) which was developed for adults who have knee OA or knee injuries.KOOS holds five subscales: (1) Pain (9 items); (2) other Symptoms (7 items); (3) Activities of Daily Living (ADL, 17 items); (4) Sport and Recreation function (Sport/Rec, 5 items); and (5) knee-related Quality of Life (QoL, 4 items). Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems)
the scale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | up to 12 months
  the WOMAC score is a disease-specific self-report multidimensional questionnare assesing pain, siffness, and physical functional disability.WOMAC scores range from 0 to 100, with higher scores indicating worse physical function.
The International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC). | up to 12 months
  The IKDC is a questionnaire that has high reliability and validity for patients with a meniscal tear. The questionnaire contains 18 items scored in 1 of 3 ways: 11-point Likert scale, 5-point Likert scale, or dichotomous yes or no. After the participant completes the questionnaire, the scores are summed, and the total score is transformed to a value on a scale of 0 to 100, with 100 representing the highest knee function.
The WOMET score | up to 12 months
  The WOMET is a meniscus-specific health-related quality-of-life instrument, validated especially for patients with a degenerative meniscal tear.The Western Ontario Meniscal Evaluation Tool (WOMET) contains 16 items addressing three domains: 9 items ad-dressing physical symptoms; 4 items addressing disabilities with regard to sports, recreation, work, and lifestyle; and 3 items addressing emotions. The score indicates the percentage of a normal score; therefore, 100 is the best possi- ble score, and 0 is the worst possible score.
height | up to 12 months
  height in meters
weight | up to 12 months
  weight in kilograms
BMI | up to 12 months
  BMI, calculated as weight in kilograms divided by height in meters squaredBMI in kg/m^2
waist circumstance | up to 12 months
  waist circumstance in centimeter
Kellgren-Lawrence grade | up to 12 months
  A Kellgren-Lawrence grade of 0 indicates no osteoarthritis, a grade of 1 with questionable osteophyte indicates possible osteoarthritis; a grade of 2 with definite osteophyte and no joint-space narrowing indicates mild osteoarthritis, a grade of 3 with ≤50% joint-space narrowing or a grade of 4 with>50% joint-space narrowing indicates severe osteoarthritis were excluded.
systolic blood pressure | up to 12 months
  systolic blood pressure in mm Hg
diastolic blood pressure | up to 12 months
  diastolic blood pressure in mm Hg
triglyceride | up to 12 months
  triglyceride in mmol/L
HDL-C | up to 12 months
  high-density lipoprotein cholesterol in mmol/L
LDL-C | up to 12 months
  low-density lipoprotein cholesterol in mmol/L
fast blood glucose | up to 12 months
  fast blood glucose in mmol/L
total Cholesterol | up to 12 months
  total Cholesterol in mmol/L
β-2 microglobulin | up to 12 months
  β-2 microglobulin in mg/L
diabetes history | up to 12 months
  diabetes history
cardio vascular disease history | up to 12 months
  cardio vascular disease history
hypertension history | up to 12 months
  hypertension history
Lysholm knee score | up to 12 months
  The Lysholm knee score is based on an eight-item questionnaire designed to evaluate knee function and symptoms in activities of daily living. Scores range from 0 to 100; higher scores indicate less severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Wang, Doctor, Principal Investigator — The First People's Hospital of Jingzhou
Locations (1):
- First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided